CLINICAL TRIAL: NCT00925509
Title: Application of Medical Imaging Procedures in Surgery Implanting in Cancerology With the Aim to Reduce Invasive Acts
Acronym: ATIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment, too much selective inclusion criteria, feasibility problems
Sponsor: Centre Leon Berard (Other)
Collaborators: French Academic Institution, Financial support: PHRC 2007 (Unknown)
Responsible Party: Centre Leon BERARD, Unité de Biostatistiques et Evaluation des Thérapeutiques
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ET2006-032; CPP 07/033 [UBET83]
Record Dates: First submitted 2009-06-02; First posted 2009-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Upper Digestive Tract Cancer
Keywords: upper digestive tract cancer; implants; implants insertion; radio-surgical guidance; accuracy of implants insertion; cranial/facial radiotherapy or brachytherapy and/or microvascular fibula transfer.; Bone volume sufficient to support an implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Therapeutic assessment -Radio-surgical guidance. — The first steps of the procedure include the production of a radiosurgical guide and the preparation of a mask in order to allow precise, non invasive repositioning of the guide.
  Secondarily, the patient undergoes a CT-scan with the mask on and the radiosurgical guide in place. This provisional scan is used for preimplantation evaluation and drilling of the guide hole.
  Under general anaesthesia, the mask is placed on the patient and the guide is fixed to the mask. A hole is drilled with a burr in the mandible through the hole in the guide. Implants are placed and the guide and mask are removed.
  A second, post-implantation CT-scan is planned 3 months after implantation. Comparison of pre- and post-implantation CT-scans allows to evaluate the precision of the placement.

SUMMARY:
Aero digestive Cancer patients treated by external head and neck radiotherapy and/or by curie-therapy and/or mandible reconstruction by microanastomosed fibula flaps. The purpose of the study is to Investigate the accuracy of implants insertion in the anteroposterior way, using radiosurgical guidance.

DETAILED DESCRIPTION:
* Investigate the accuracy of inserting implants in the vertical way and in angulation, on irradiated native mandible or on microanastomosed fibula flaps
* Investigate the accuracy of inserting implants in the anteroposterior way, in the vertical way and in angulation for all the involved patients (meaning on irradiated native mandible or on microanastomosed fibula flaps)
* Investigate the delay of mucous healing
* Estimate the prosthetic function
* Evaluate the osteonecrosis rate after radiation with traumatic etiology due to implantation
* Estimate the implant rate due to minimally invasive flaps
* Estimate the implant rate due to pure trans mucosa way
* Estimate the post surgical therapeutic success after 1 year

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* Performance status over 70
* Histological evidence of upper digestive tract cancer
* History of cranial / facial radiotherapy or brachytherapy and/or microvascular fibula transfer.
* Bone volume sufficient to support an implant.
* Mandatory affiliation with a social security system
* Written, voluntary, informed consent

Exclusion Criteria:

* Patient with evolutive malignant disease
* Contraindication to general anesthesia
* Concurrent disease contra-indicating implant surgery (risk of infectious endocarditis, uncontrolled diabetes, HIV, evolutive neoplasia…)
* Patient enrolled in another clinical trial including chemotherapy
* Pregnant or lactating woman
* Anticipation of an impossible follow-up
* Patient deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of implants insertion, radio-surgical guidance. | 8 months after inclusion

SECONDARY OUTCOMES:
Accuracy of inserting implants | 16 months after inclusion
Delay of mucous healing | 16 months after inclusion
Estimation of the prosthetic function | 16 months after inclusion
Osteonecrosis rate after radiation with traumatic etiology due to implantation | 16 months after inclusion
Implant rate | 16 months after inclusion
Post surgical therapeutic success after 1 year | after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Gaëlle BODARD, MD, Principal Investigator — Centre Leon Berard
Locations (4):
- France (4):
  - Centre Léon Bérard Service de Chirurgie-Stomatologie, Lyon, Cedex 08
  - CHU Hôtel-Dieu Service d'Odontologie, Clermont-Ferrand
  - Hospices Civils de Lyon Service de Consultations et Traitements Dentaires, Lyon
  - Centre Hospitalier Lyon Sud Service de Stomatologie et Chirurgie Maxillo-Faciale, Pierre-Bénite

REFERENCES:
- [Background] Beumer J 3rd, Roumanas E, Nishimura R. Advances in osseointegrated implants for dental and facial rehabilitation following major head and neck surgery. Semin Surg Oncol. 1995 May-Jun;11(3):200-7. doi: 10.1002/ssu.2980110305. PMID 7638507
- [Background] Birkfellner W, Solar P, Gahleitner A, Huber K, Kainberger F, Kettenbach J, Homolka P, Diemling M, Watzek G, Bergmann H. In-vitro assessment of a registration protocol for image guided implant dentistry. Clin Oral Implants Res. 2001 Feb;12(1):69-78. doi: 10.1034/j.1600-0501.2001.012001069.x. PMID 11168273
- [Background] Brosky ME, Korioth TW, Hodges J. The anterior cantilever in the implant-supported screw-retained mandibular prosthesis. J Prosthet Dent. 2003 Mar;89(3):244-9. doi: 10.1067/mpr.2003.43. PMID 12644798
- [Background] Casap N, Wexler A, Persky N, Schneider A, Lustmann J. Navigation surgery for dental implants: assessment of accuracy of the image guided implantology system. J Oral Maxillofac Surg. 2004 Sep;62(9 Suppl 2):116-9. doi: 10.1016/j.joms.2004.06.028. PMID 15332188
- [Background] Casap N, Wexler A, Tarazi E. Application of a surgical navigation system for implant surgery in a deficient alveolar ridge postexcision of an odontogenic myxoma. J Oral Maxillofac Surg. 2005 Jul;63(7):982-8. doi: 10.1016/j.joms.2005.03.015. PMID 16003627
- [Background] Delannes M, Daly NJ, Bonnet J, Sabatier J, Tremoulet M. Fractionated radiotherapy of small inoperable lesions of the brain using a non-invasive stereotactic frame. Int J Radiat Oncol Biol Phys. 1991 Aug;21(3):749-55. doi: 10.1016/0360-3016(91)90695-z. PMID 1869468
- [Background] Esser E, Wagner W. Dental implants following radical oral cancer surgery and adjuvant radiotherapy. Int J Oral Maxillofac Implants. 1997 Jul-Aug;12(4):552-7. PMID 9274085
- [Background] Esser E, Neukirchen S, Wagner W. [Comparative studies of Branemark implants in the irradiated and not irradiated mandible]. Mund Kiefer Gesichtschir. 1999 May;3 Suppl 1:S125-9. doi: 10.1007/PL00014498. German. PMID 10414098
- [Background] Fortin T, Coudert JL, Champleboux G, Sautot P, Lavallee S. Computer-assisted dental implant surgery using computed tomography. J Image Guid Surg. 1995;1(1):53-8. doi: 10.1002/(SICI)1522-712X(1995)1:13.0.CO;2-L. PMID 9079427
- [Background] Fortin T, Champleboux G, Lormee J, Coudert JL. Precise dental implant placement in bone using surgical guides in conjunction with medical imaging techniques. J Oral Implantol. 2000;26(4):300-3. doi: 10.1563/1548-1336(2000)0262.3.CO;2. PMID 11831236
- [Background] Fortin T, Champleboux G, Bianchi S, Buatois H, Coudert JL. Precision of transfer of preoperative planning for oral implants based on cone-beam CT-scan images through a robotic drilling machine. Clin Oral Implants Res. 2002 Dec;13(6):651-6. doi: 10.1034/j.1600-0501.2002.130612.x. PMID 12519341
- [Background] Fortin T, Bosson JL, Coudert JL, Isidori M. Reliability of preoperative planning of an image-guided system for oral implant placement based on 3-dimensional images: an in vivo study. Int J Oral Maxillofac Implants. 2003 Nov-Dec;18(6):886-93. PMID 14696665
- [Background] Fortin T, Isidori M, Blanchet E, Perriat M, Bouchet H, Coudert JL. An image-guided system-drilled surgical template and trephine guide pin to make treatment of completely edentulous patients easier: a clinical report on immediate loading. Clin Implant Dent Relat Res. 2004;6(2):111-9. doi: 10.1111/j.1708-8208.2004.tb00033.x. PMID 15669711
- [Background] Ganslandt O, Mueller R, Mueller W, Borchert H, Grabenbauer GG. Simple invasive fixation device for fractionated stereotactic LINAC based radiotherapy. Acta Neurochir (Wien). 2003 Apr;145(4):289-94; discussion 294. doi: 10.1007/s00701-003-0002-9. PMID 12748889
- [Background] Gill SS, Thomas DG, Warrington AP, Brada M. Relocatable frame for stereotactic external beam radiotherapy. Int J Radiat Oncol Biol Phys. 1991 Mar;20(3):599-603. doi: 10.1016/0360-3016(91)90076-g. PMID 1995547
- [Background] Gulizio MP, Agar JR, Kelly JR, Taylor TD. Effect of implant angulation upon retention of overdenture attachments. J Prosthodont. 2005 Mar;14(1):3-11. doi: 10.1111/j.1532-849X.2005.00005.x. PMID 15733129
- [Background] Henderson LA, Frysinger RC, Yu PL, Bandler R, Harper RM. A device for feline head positioning and stabilization during magnetic resonance imaging. Magn Reson Imaging. 2001 Sep;19(7):1031-6. doi: 10.1016/s0730-725x(01)00423-4. PMID 11595376
- [Background] Kamath R, Ryken TC, Meeks SL, Pennington EC, Ritchie J, Buatti JM. Initial clinical experience with frameless radiosurgery for patients with intracranial metastases. Int J Radiat Oncol Biol Phys. 2005 Apr 1;61(5):1467-72. doi: 10.1016/j.ijrobp.2004.08.021. PMID 15817352
- [Background] Kassaee A, Das IJ, Tochner Z, Rosenthal DI. Modification of Gill-Thomas-Cosman frame for extracranial head-and-neck stereotactic radiotherapy. Int J Radiat Oncol Biol Phys. 2003 Nov 15;57(4):1192-5. doi: 10.1016/s0360-3016(03)00774-0. PMID 14575852
- [Background] Marunick MT, Leveque F. Osteoradionecrosis related to mastication and parafunction. Oral Surg Oral Med Oral Pathol. 1989 Nov;68(5):582-5. doi: 10.1016/0030-4220(89)90244-2. PMID 2812713
- [Background] Medin PM, Solberg TD, De Salles AA, Cagnon CH, Selch MT, Johnson JP, Smathers JB, Cosman ER. Investigations of a minimally invasive method for treatment of spinal malignancies with LINAC stereotactic radiation therapy: accuracy and animal studies. Int J Radiat Oncol Biol Phys. 2002 Mar 15;52(4):1111-22. doi: 10.1016/s0360-3016(01)02762-6. PMID 11958909
- [Background] Parel SM, Triplett RG. Interactive imaging for implant planning, placement, and prosthesis construction. J Oral Maxillofac Surg. 2004 Sep;62(9 Suppl 2):41-7. doi: 10.1016/j.joms.2004.05.207. PMID 15332180
- [Background] Quinones-Hinojosa A, Ware ML, Sanai N, McDermott MW. Assessment of image guided accuracy in a skull model: comparison of frameless stereotaxy techniques vs. frame-based localization. J Neurooncol. 2006 Jan;76(1):65-70. doi: 10.1007/s11060-005-2915-z. PMID 16132501
- [Background] Rosenberg I, Alheit H, Beardmore C, Lee KS, Warrington AP, Brada M. Patient position reproducibility in fractionated stereotactic radiotherapy: an update after changing dental impression material. Radiother Oncol. 1999 Feb;50(2):239-40. doi: 10.1016/s0167-8140(99)00002-x. PMID 10368049
- [Background] Rosenthal SJ, Gall KP, Jackson M, Thornton AF Jr. A precision cranial immobilization system for conformal stereotactic fractionated radiation therapy. Int J Radiat Oncol Biol Phys. 1995 Dec 1;33(5):1239-45. doi: 10.1016/0360-3016(95)02009-8. PMID 7493848
- [Background] Scott TW, Beach JL, Mendiondo OA. A precision repeat localization head frame for fractionated stereotactic radiotherapy. Med Dosim. 1997 Spring;22(1):5-8. doi: 10.1016/s0958-3947(96)00148-3. PMID 9136100
- [Background] Siessegger M, Schneider BT, Mischkowski RA, Lazar F, Krug B, Klesper B, Zoller JE. Use of an image-guided navigation system in dental implant surgery in anatomically complex operation sites. J Craniomaxillofac Surg. 2001 Oct;29(5):276-81. doi: 10.1054/jcms.2001.0242. PMID 11673922
- [Background] Sudbrink SD. Computer-guided implant placement with immediate provisionalization: a case report. J Oral Maxillofac Surg. 2005 Jun;63(6):771-4. doi: 10.1016/j.joms.2005.02.011. PMID 15944973
- [Background] Theodorou K, Kappas C, Tsokas C. A new non-invasive and relocatable immobilization frame for fractionated stereotactic radiotherapy. Radiother Oncol. 1998 Jun;47(3):313-7. doi: 10.1016/s0167-8140(98)00015-2. PMID 9681896
- [Background] Van Steenberghe D, Malevez C, Van Cleynenbreugel J, Bou Serhal C, Dhoore E, Schutyser F, Suetens P, Jacobs R. Accuracy of drilling guides for transfer from three-dimensional CT-based planning to placement of zygoma implants in human cadavers. Clin Oral Implants Res. 2003 Feb;14(1):131-6. doi: 10.1034/j.1600-0501.2003.140118.x. PMID 12562376
- [Background] Vrielinck L, Politis C, Schepers S, Pauwels M, Naert I. Image-based planning and clinical validation of zygoma and pterygoid implant placement in patients with severe bone atrophy using customized drill guides. Preliminary results from a prospective clinical follow-up study. Int J Oral Maxillofac Surg. 2003 Feb;32(1):7-14. doi: 10.1054/ijom.2002.0337. PMID 12653226
- [Background] Wagner A, Wanschitz F, Birkfellner W, Zauza K, Klug C, Schicho K, Kainberger F, Czerny C, Bergmann H, Ewers R. Computer-aided placement of endosseous oral implants in patients after ablative tumour surgery: assessment of accuracy. Clin Oral Implants Res. 2003 Jun;14(3):340-8. doi: 10.1034/j.1600-0501.2003.110812.x. PMID 12755784
- [Background] Watzinger F, Ewers R, Henninger A, Sudasch G, Babka A, Woelfl G. Endosteal implants in the irradiated lower jaw. J Craniomaxillofac Surg. 1996 Aug;24(4):237-44. doi: 10.1016/s1010-5182(96)80007-2. PMID 8880450
- [Background] Weischer T, Schettler D, Mohr C. Implant-supported telescopic restorations in maxillofacial prosthetics. Int J Prosthodont. 1997 May-Jun;10(3):287-92. PMID 9484062
- [Background] Weischer T, Mohr C. Ten-year experience in oral implant rehabilitation of cancer patients: treatment concept and proposed criteria for success. Int J Oral Maxillofac Implants. 1999 Jul-Aug;14(4):521-8. PMID 10453667
- [Background] Weischer T, Mohr C. Implant-supported mandibular telescopic prostheses in oral cancer patients: an up to 9-year retrospective study. Int J Prosthodont. 2001 Jul-Aug;14(4):329-34. PMID 11508087
- [Background] Widmann G, Widmann R, Widmann E, Jaschke W, Bale RJ. In vitro accuracy of a novel registration and targeting technique for image-guided template production. Clin Oral Implants Res. 2005 Aug;16(4):502-8. doi: 10.1111/j.1600-0501.2005.01131.x. PMID 16117777
- [Background] Kooy HM, Dunbar SF, Tarbell NJ, Mannarino E, Ferarro N, Shusterman S, Bellerive M, Finn L, McDonough CV, Loeffler JS. Adaptation and verification of the relocatable Gill-Thomas-Cosman frame in stereotactic radiotherapy. Int J Radiat Oncol Biol Phys. 1994 Oct 15;30(3):685-91. doi: 10.1016/0360-3016(92)90956-i. PMID 7928501